CLINICAL TRIAL: NCT00258830
Title: Annual Study of Safety and Immunogenicity of Fluzone® Influenza Virus Vaccine (2005-2006 Formulation)
Brief Title: Safety and Immunogenicity of the 2005-2006 Fluzone® Vaccine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GRC25
Record Dates: First submitted 2005-11-24; First posted 2005-11-28 (Estimated); Results first posted 2009-06-03 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2016-04

CONDITIONS: Influenza
Keywords: Influenza vaccine
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Age 18 to 59 years (Experimental): Participants aged 18 to 59 years at enrollment.
  Interventions: Biological: Fluzone®: Influenza Virus Vaccine
- Age 60 years and older (Experimental): Participants aged 60 years and older at enrollment.
  Interventions: Biological: Fluzone®: Influenza Virus Vaccine

INTERVENTIONS:
Biological: Fluzone®: Influenza Virus Vaccine — 0.5 mL, Intramuscular
  Other Names: Fluzone®
  Arms: Age 18 to 59 years
Biological: Fluzone®: Influenza Virus Vaccine — 0.5 mL, Intramuscular
  Other Names: Fluzone®
  Arms: Age 60 years and older

SUMMARY:
To describe the safety during Days 0 to 21 following injection of the 2005-2006 formulation of the inactivated, split-virion influenza vaccine Fluzone in subjects aged 18-59 years and subjects aged ≥ 60 years.

To describe the immune response (antibodies to hemagglutinin) 21 days following injection of the 2005-2006 formulation of the inactivated, split-virion influenza vaccine Fluzone, in subjects aged 18-59 years and subjects aged ≥ 60 years.

To submit remaining available sera to the Center for Biologics Evaluation and Research (CBER) for further analysis by the Food and Drug Administration (FDA), Center for Disease Control and Prevention (CDC) and the World Health Organization (WHO) to support selection and recommendation of antigen strains for subsequent influenza vaccines.

ELIGIBILITY:
Inclusion Criteria:

* Participant aged 18 years or older on the day of inclusion.
* Participant able to attend scheduled visits and to comply with the study procedures during the entire duration of the study.
* Participant is in reasonably good health as assessed by the investigator.
* Participant willing and able to meet protocol requirements.
* Participant willing and able to give informed consent.
* For a woman, inability to bear a child or negative serum/urine pregnancy test.

Exclusion Criteria:

* Self-reported allergy to egg proteins, chicken proteins, or one of the constituents of the vaccine, such as thimerosal or formaldehyde.
* An acute illness with or without fever (temperature ≥ 99.5°F oral) in the 72 hours preceding enrollment in the trial.
* Clinically significant findings in vital signs (including temperature ≥ 99.5°F oral) on review of systems.
* Self-reported history of severe adverse event to any influenza vaccine.
* Laboratory-confirmed influenza infection or vaccination against influenza in the 6 months preceding enrollment in the study.
* Any vaccination in the 14 days preceding enrollment in the study or scheduled between Visit 1 and Visit 3.
* Vaccination planned in the 4 weeks following any trial vaccination.
* Participation in any other interventional drug or vaccine trial within the 30 days preceding or during enrollment into this study.
* Immunocompromising or immunosuppressive therapy (including systemic steroid use for 2 weeks or more), cancer chemotherapy, or radiation therapy at the time of enrollment, planned during the period of this study, or at any time within the past 6 months.
* Receipt of blood or blood products within the 3 months preceding enrollment in the study.
* Diabetes mellitus requiring pharmacological control.
* Any condition that in the opinion of the Investigator posed a health risk to the subject if enrolled or interfered with the evaluation of the vaccine.
* Person deprived of freedom by an administrative or court order (having legal or medical guardian).
* For women of childbearing potential, a positive urine pregnancy test, breast feeding, or not using a medically approved form of contraception for the duration of the trial.
* Current abuse of alcohol or drug addiction that interfered with the subject's ability to comply with trial procedures.
* Thrombocytopenia or bleeding disorder contraindicating intramuscular (IM) vaccination.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2005-09; Primary Completion 2006-02 (Actual); Study Completion 2007-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc.
Locations (1):
- Norfolk, Virginia, United States

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants were enrolled from 09 September to 18 October 2005 in one medical clinic in the US
Pre-assignment Details: A total of 120 subjects that met the inclusion and exclusion criteria were enrolled and vaccinated.
Groups:
- Age 18 to 59 Years: Participants aged 18 to 59 years at enrollment received 0.5 mL of Fluzone® vaccine intramuscularly.
- Age 60 Years and Older: Participants aged 60 years and older at enrollment received 0.5 mL of Fluzone® vaccine intramuscularly.
Period: Overall Study
Arm/Group | Age 18 to 59 Years | Age 60 Years and Older
Started | 60 | 60
Completed | 60 | 60
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Age 18 to 59 Years | Age 60 Years and Older | Total
Number analyzed (Participants) | 60 | 60 | 120
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 0 | 1
  Between 18 and 65 years | 59 | 2 | 61
  >=65 years | 0 | 58 | 58
Age, Continuous [Mean (Standard Deviation); unit: Years] | 42.8 (11.25) | 75.7 (6.24) | 59.3 (18.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 39 | 88
  Male | 11 | 21 | 32
Region of Enrollment [Number; unit: participants]
  United States | 60 | 60 | 120

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting Solicited Injection Site and Solicited Systemic Reactions After Fluzone® Vaccination
Time Frame: Day 0 to 3 post-vaccination
Population: Safety analysis was on all enrolled and vaccinated subjects intent-to-treat safety population with available reaction data.
Measure: Number; unit: Participants
Arm/Group | Age 18 to 59 Years | Age 60 Years and Older
Number analyzed (Participants) | 60 | 60
Participants
  Any Solicited Injection Site Reaction | 40 | 10
  Any Erythema | 4 | 6
  Grade 3 Erythema (≥ 5.0 cm) | 1 | 1
  Any Swelling | 3 | 3
  Grade 3 Swelling (≥ 5.0 cm) | 1 | 0
  Any Pain | 39 | 8
  Grade 3 Pain (Unable to perform usual activities) | 0 | 0
  Any Solicited Systemic Reaction | 25 | 9
  Any Fever | 0 | 2
  Grade 3 Fever (≥ 102.3°F) | 0 | 0
  Any Headache | 12 | 3
  Grade 3 Headache (Prevents daily activity) | 1 | 0
  Any Malaise | 7 | 4
  Grade 3 Malaise (Prevents daily activity) | 0 | 0
  Any Myalgia | 13 | 3
  Grade 3 Myalgia (Prevents daily activity) | 0 | 0

2. Primary Outcome: Geometric Mean Titers (GMTs) of Hemagglutination Antibodies Before and After Fluzone® Vaccination
Description: GMTs and their 95% Confidence Intervals are presented for each of the 3 antigens in Fluzone® vaccine (2005-2006 Formulation)
Time Frame: 21 days post-vaccination
Population: GMT results were assessed on the per-protocol population.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Age 18 to 59 Years | Age 60 Years and Older
Number analyzed (Participants) | 60 | 60
Titer
  A/New Caledonia/20/99 (H1N1), Pre | 51.8 [35.9 to 74.8] | 34.8 [27.7 to 43.8]
  A/New Caledonia/20/99 (H1N1), Post | 153.6 [113.8 to 207.2] | 59.3 [45.9 to 76.6]
  A/New York/55/2004 (H3N2), Pre | 23.9 [18.2 to 31.5] | 23.1 [16.8 to 31.9]
  A/New York/55/2004 (H3N2), Post | 341.0 [241.0 to 482.5] | 174.5 [116.8 to 260.7]
  B/Jiangsu/10/2003, Pre | 25.9 [19.4 to 34.6] | 42.6 [33.3 to 54.6]
  B/Jiangsu/10/2003, Post | 126.5 [93.0 to 172.1] | 104.8 [78.3 to 140.4]

3. Other Pre Specified Outcome: Percentage of Participants With ≥ 40 Serum Hemagglutination Inhibition Antibody Titers Post-vaccination.
Description: Seroprotection: Percentage of participants with ≥ 40 serum hemagglutination inhibition antibody titers 21 days post-vaccination.
Time Frame: 21 Days post-vaccination
Population: Seroprotection was assessed in the per-protocol population
Measure: Number; unit: Percentage of participants
Arm/Group | Age 18 to 59 Years | Age 60 Years and Older
Number analyzed (Participants) | 60 | 60
Percentage of participants
  A/New Caledonia/20/99 (H1N1) ≥ 40 | 90 | 71
  A/New York/55/2004 (H3N2) ≥ 40 | 95 | 83
  B/Jiangsu/10/2003 ≥ 40 | 86 | 83

4. Other Pre Specified Outcome: Percentage of Participants With a ≥ 4-fold Increase in Serum Hemagglutination Inhibition Antibody Titers Post-vaccination
Description: Seroconversion: percentage of participants with at least a 4-fold increase in serum hemagglutination inhibition antibody titers at 21 days post-vaccination.
Time Frame: Day 21 post-vaccination
Population: Seroconversion was assessed in the per-protocol population.
Measure: Number; unit: Percentage of participants
Arm/Group | Age 18 to 59 Years | Age 60 Years and Older
Number analyzed (Participants) | 60 | 60
Percentage of participants
  A/New Caledonia/20/99 (H1N1) ≥ 4 fold-rise | 29 | 9
  A/New York/55/2004 (H3N2) ≥ 4 fold-rise | 93 | 67
  B/Jiangsu/10/2003 ≥ 4 fold-rise | 54 | 27

ADVERSE EVENTS:
Time Frame: Adverse events data were collected from the day of vaccination for 28 days post-vaccination.
Arm/Group | Age 18 to 59 Years | Age 60 Years and Older
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/60
Other Adverse Events (participants affected / at risk) | 15/60 | 5/60
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Age 18 to 59 Years (N=60) | Age 60 Years and Older (N=60)
Nasopharyngitis (Infections and infestations) | 0 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 0
Headache (Nervous system disorders) | 12 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.